CLINICAL TRIAL: NCT04653402
Title: Determine the Efficacy of Closed Suction Drain After Hydrocelectomy in Primary Vaginal Hydrocele: An Open-label Randomised Controlled Trial (END Trial)
Brief Title: Determine the Efficacy of Closed Suction Drain After Hydrocelectomy. (END Trial)
Acronym: END
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Prakash Kumar Sasmal, Additional Professor,Dept of General Surgery, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T/IM-NF/Gen.Surg/20/45
Record Dates: First submitted 2020-10-10; First posted 2020-12-04 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Hydrocele of Tunica Vaginalis
Keywords: Hydrocele; Drain; Surgery; Complications; Hydrocelectomy; Hematoma; Infection
MeSH Terms: conditions — Testicular Hydrocele; Hematoma; Infections

STUDY DESIGN:
Intervention Model Description: open label randomised control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study arm 1 (Experimental): Placing a closed suction drain after hydrocelectomy for primary vaginal hydrocele
  Interventions: Device: Hydrocelectomy surgery
- Study arm 2 (Active Comparator): Not placing a drain after hydrocelectomy in primary vaginal hydrocele
  Interventions: Device: Hydrocelectomy surgery

INTERVENTIONS:
Device: Hydrocelectomy surgery — The standardized hydrocelectomy operation i.e. Eversion of the TVT sac

SUMMARY:
There is no clear consensus regarding the benefits of putting a closed suction drain after eversion of the sac in a hydrocele of the tunica vaginalis testis. Our study will find out the benefits if at all of a closed suction drain in hydrocele surgery. The potential complications expected after hydrocelectomy surgery are bleeding, infection, redness, and pain. There is no such trial to date to determine the benefits of putting a closed suction drain after hydrocelectomy surgery.

DETAILED DESCRIPTION:
Study objectives:

1. Primary:

   To compare the postoperative complication rates of hematoma, skin edema and surgical site infection after hydrocelectomy, between patients with or without a closed suction drain (CSD).
2. Secondary:

To compare postoperative pain (testalgia) between the two groups of patients.

Study setting: All patients over 18 years of age attending the outpatient department of General Surgery at AIIMS, Bhubaneswar with the diagnosis of idiopathic hydrocele and planned for elective surgery.

Total Sample Size = 60 (30 in each arm)

ELIGIBILITY:
Inclusion Criteria:

- All patients over 18 years of age diagnosed with primary hydrocele by clinical and ultrasonographic confirmation, undergoing hydrocelectomy surgery.

Exclusion Criteria:

* Patient not giving consent to participate
* Patients with ASA (American Society of Anaesthesiology) grade 3 & 4
* Patients with congenital or secondary hydrocele
* Patients with recurrent disease, pyocele or filarial scrotum

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Skin edema | Post operative period of 1 month
  Boggy swelling of scrotal wall
Hematoma | Post operative period of 1 month
  Post-operative swelling of scrotum with skin discolouration and oozing of blood through the incision site
Surgical site infection | Post operative period of 1 month
  Seropurulent discharge from the incision site with systemic signs of infection like fever, tachycardia and local signs like edema, redness and tenderness

SECONDARY OUTCOMES:
Testalgia | post operative period of 1 month
  Visual Analog Scale scoring on a 100 mm length scale ( low score with no pain to higher scores with worst imaginable pain) for acute and sub acute testalgia

CONTACTS AND LOCATIONS:
Overall Officials: Prakash K. Sasmal, MS,FNB,FAIS, Principal Investigator — All India Institute of Medical Sciences, Bhubaneswar, INDIA
Locations (1):
- All India institute of medical sciences, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: Yes
Participant information sheet and participant consent form and study protocol.
Supporting Information: Study Protocol, ICF
Time Frame: Before the start of the study
Access Criteria: IEC

REFERENCES:
- [Background] Dagur G, Gandhi J, Suh Y, Weissbart S, Sheynkin YR, Smith NL, Joshi G, Khan SA. Classifying Hydroceles of the Pelvis and Groin: An Overview of Etiology, Secondary Complications, Evaluation, and Management. Curr Urol. 2017 Apr;10(1):1-14. doi: 10.1159/000447145. Epub 2017 Mar 30. PMID 28559772
- [Background] Tsai L, Milburn PA, Cecil CL 4th, Lowry PS, Hermans MR. Comparison of Recurrence and Postoperative Complications Between 3 Different Techniques for Surgical Repair of Idiopathic Hydrocele. Urology. 2019 Mar;125:239-242. doi: 10.1016/j.urology.2018.12.004. Epub 2018 Dec 12. PMID 30552941
- [Background] Agbakwuru EA, Salako AA, Olajide AO, Takure AO, Eziyi AK. Hydrocelectomy under local anaesthesia in a Nigerian adult population. Afr Health Sci. 2008 Sep;8(3):160-2. PMID 19357743
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Result] Patil V, Shetty SM, Das S. Common and Uncommon Presentation of Fluid within the Scrotal Spaces. Ultrasound Int Open. 2015 Nov;1(2):E34-40. doi: 10.1055/s-0035-1555919. Epub 2015 Nov 6. PMID 27689151
- See also: Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. — https://pubmed.ncbi.nlm.nih.gov/26092476/
- See also: Hydrocelectomy under local anaesthesia in a Nigerian adult population. — https://pubmed.ncbi.nlm.nih.gov/19357743/
- See also: omparison of Recurrence and Postoperative Complications Between 3 Different Techniques for Surgical Repair of Idiopathic Hydrocele. — http://pubmed.ncbi.nlm.nih.gov/30552941
- See also: Common and Uncommon Presentation of Fluid within the Scrotal Spaces. Ultrasound Int Open — http://pubmed.ncbi.nlm.nih.gov/27689151/